CLINICAL TRIAL: NCT00475254
Title: Stress and Vision Fluctuations in Retinitis Pigmentosa
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Ava Bittner, OD, PhD, Johns Hopkins University
Other Study IDs: K23EY018356 (NIH)
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2008-08

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; stress; sleepiness; low vision; mind-body
MeSH Terms: conditions — Retinitis Pigmentosa; Sleepiness; Vision, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Retinitis pigmentosa (RP) patients experience a slowly progressive, unpredictable loss of vision which eventually leads to bare or no light perception, posing a continuous threat to patients' independence. Negative psychological states such as distress, sleepiness, anxiety and depression are common in RP patients due to the nature of this chronic, disabling disease. Psychophysical vision measures are more variable in legally blind RP subjects than in normally sighted individuals, and RP patients indicate that variations in vision are often related to stress. The primary goal of this research is to examine the vision fluctuations within and between days among RP patients using vision tests self-administered by patients through their home computers, and determine associations with factors such as perceived stress, mood states, sleepiness, or light exposure. The administration of questionnaires will allow us to gain some insight into which underlying psychological factors impact certain vision measures, allowing the design of future interventional research to attempt to reduce such factors. The aims of many future treatment clinical trials for RP will be to improve vision and/or reduce the rate of vision loss; thus the sources that lead to increased variability of vision need to be identified and alleviated to enable precise evaluation of interventions and improve patients' quality of life.

DETAILED DESCRIPTION:
An initial study visit for enrollment will take place at the Johns Hopkins Wilmer Eye Institute's Lions Vision Center. The investigators will enroll 50 RP subjects with vision better than hand motions or bare light perception, who are able to complete PC-based vision tests. Written informed consent for study participation will be obtained at the first study visit.

At home PC-based vision tests will be performed bi-weekly, for 2 months (i.e. 16 measures) to capture the full range of variability. Binocular visual acuity (VA), contrast sensitivity (CS) and visual field (VF) tests will be self-administered by the RP subjects, and will take ~10 minutes. Three brief questionnaires will be administered by PC after each vision test session: 1) Perceived Stress Scale (PSS); 2) Stanford Sleepiness Scale (SSS); and 3) Positive and Negative Affect Schedules (PANAS). Lab-based vision tests will take place at the time of enrollment, and will include: (1) distance best-corrected VA with the ETDRS charts, (2) Pelli-Robson letter CS, (3) Goldmann VF with V/4e and III/4e isopters, and (4) Humphrey 10-2 or 30-2 VF FastPac program. The vision tests and questionnaires are a part of routine clinical care.

After enrollment, The investigators will obtain information about psychological factors by administering the following questionnaires by phone on one occasion: Pittsburgh Sleep Quality Index, Emotional Stability, Beck Depression Inventory, the Self-Motivation Inventory, and the Life Experiences Survey. Questionnaires assessing health-related quality of life (SF-36) and mental status (MMSE) will also be administered. The investigators will use a phone version of the MMSE only for screening. Other variables that may be of importance to the study will be assessed through a complete patient medical, ocular and social history, including questions such as duration of visual impairment, occupation, marital status, etc. The questionnaires are often used in research settings and sometimes in clinical settings. Many patients appreciate the opportunity to provide feedback since these areas are not always addressed as part of routine, clinical care. Focus group meetings, facilitated by Dr. George and Lori Edwards, will help us begin to understand factors are perceived to influence fluctuations in vision.

Subjects will participate in study procedures over the course of a 3 month period. This includes an enrollment visit at our center with lab-based vision tests, and then approximately 2 months PC-based vision testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed retinitis pigmentosa

Exclusion Criteria:

* Very severe vision loss (i.e., light perception only) who may have difficulty performing the vision tests with their home computers
* Unable to use a PC (Personal Computer)
* Non-English speaking
* Unable to communicate experiences
* Out of town for more than one week during a 2 month period when taking the PC-based tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with a confirmed diagnosis of retinitis pigmentosa
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Vision test reliability across multiple test administrations in relation to psychological and external factors | 2-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ava K. Bittner, O.D., Ph.D., Principal Investigator — Johns Hopkins Wilmer Eye Institute; Maureen George, Ph.D., Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins WiImer Eye Insitute's Lions Vision Center, Baltimore, Maryland, United States

REFERENCES:
- See also: Johns Hopkins Center for Mind-Body Research — http://www.jhsph.edu/mindbodyresearch/